CLINICAL TRIAL: NCT02288143
Title: Evaluation of a Simplified Low-cost and Friendly Controlled Ovarian Stimulation Combining Oral Letrozole and Clomiphene Citrate: a Pilot Study
Brief Title: COmbining Oral Letrozole and Clomiphene for Ovarian Stimulation
Acronym: COOL-COS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Wellington P Martins, MD, Associate Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 37537014.6.0000.5440
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COOL-COS (Experimental): All women will receive the intervention: Letrozole, Clomiphene, and low-dose hMG for the controlled ovarian stimulation.
  Interventions: Drug: COOL-COS

INTERVENTIONS:
Drug: COOL-COS — Controlled ovarian stimulation will start on the second or third day of a menstrual cycle:
  * Oral clomiphene citrate: 100 mg/day until the day of the triggering.
  * Oral letrozole: 7.5 mg/day during the first 5 days of the controlled ovarian stimulation.
  * hMG: 150 IU every other day beginning on the day 6 of the controlled ovarian stimulation.
  The triggering will be performed using urinary hCG (5,000 IU subcutaneous).
  * 1-2 days after the identification of one follicle ≥ 17 mm
  * 0-1 days after the identification of one follicle ≥ 19 mm.
  Other Names: Friendly COS

SUMMARY:
This is a pilot study evaluating the effect of a simplified low-cost (friendly) controlled ovarian stimulation using clomiphene citrate, letrozole, and low-dose hMG on the number of oocytes retrieved.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled to controlled ovarian stimulation for oocyte retrieval.
* Body mass index: 18-35 Kg/m2.
* Ultrasound scan up to the third day of a menstrual cycle with absence of a dominant and active follicle (follicle >10mm and serum estradiol ≥ 40 pg/L).
* Signing an informed consent.

Exclusion Criteria:

* No exclusion criteria.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 12 days

SECONDARY OUTCOMES:
Number of embryos | 17 days
Ovarian hyper-stimulation syndrome | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Setor de Reproducao Humana do HC-FMRP-USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Figueiredo JB, Nastri CO, Vieira AD, Martins WP. Clomiphene combined with gonadotropins and GnRH antagonist versus conventional controlled ovarian hyperstimulation without clomiphene in women undergoing assisted reproductive techniques: systematic review and meta-analysis. Arch Gynecol Obstet. 2013 Apr;287(4):779-90. doi: 10.1007/s00404-012-2672-0. Epub 2012 Dec 19. PMID 23250342
- [Result] Hajishafiha M, Dehghan M, Kiarang N, Sadegh-Asadi N, Shayegh SN, Ghasemi-Rad M. Combined letrozole and clomiphene versus letrozole and clomiphene alone in infertile patients with polycystic ovary syndrome. Drug Des Devel Ther. 2013 Dec 3;7:1427-31. doi: 10.2147/DDDT.S50972. eCollection 2013. PMID 24348019
- [Result] Martins WP, Vieira AD, Figueiredo JB, Nastri CO. FSH replaced by low-dose hCG in the late follicular phase versus continued FSH for assisted reproductive techniques. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD010042. doi: 10.1002/14651858.CD010042.pub2. PMID 23543584
- [Result] Seko LM, Moroni RM, Leitao VM, Teixeira DM, Nastri CO, Martins WP. Melatonin supplementation during controlled ovarian stimulation for women undergoing assisted reproductive technology: systematic review and meta-analysis of randomized controlled trials. Fertil Steril. 2014 Jan;101(1):154-161.e4. doi: 10.1016/j.fertnstert.2013.09.036. Epub 2013 Oct 29. PMID 24182414
- [Result] Nastri CO, Teixeira DM, Moroni RM, Leitao VM, Martins WP. Ovarian hyperstimulation syndrome: pathophysiology, staging, prediction and prevention. Ultrasound Obstet Gynecol. 2015 Apr;45(4):377-93. doi: 10.1002/uog.14684. Epub 2015 Mar 1. PMID 25302750